CLINICAL TRIAL: NCT00613405
Title: Stress and Marijuana Cue-elicited Craving and Reactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Aimee McRae-Clark, Associate Professor of Psychiatry, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: HR#17195; R21DA022424 (NIH); R21DA022424-01A1 (NIH)
Record Dates: First submitted 2008-02-11; First posted 2008-02-13 (Estimated); Results first posted 2012-05-04 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Cannabis Use Disorders
Keywords: substance-related disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Psychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stress + cue exposure (Experimental): Individuals were exposed to the Trier Social Stress Test (TSST) as well as neutral cues and marijana cues.
  Interventions: Other: Stress + cue exposure
- No stress + cue exposure (Experimental): Individuals were not exposed to a stress test, but were exposed to neutral cues and marijuana cues.
  Interventions: Other: No stress + cue exposure

INTERVENTIONS:
Other: Stress + cue exposure — Trier Social Stress Task(TSST): subject is asked to give a talk and perform a math task in front of an audience, follwed by neutral and marijuana cue exposure.
  Other Names: Stress stask, TSST
  Arms: Stress + cue exposure
Other: No stress + cue exposure — Neutral and marijuana-associated cue exposure (scripted imagery, in vivo cues).
  Other Names: marijuana cue exposure, neutral cue exposure
  Arms: No stress + cue exposure

SUMMARY:
The purpose of this study is to explore the interaction between stress and marijuana cues, in hopes that it may lead to the development of new treatments for marijuana dependence.

DETAILED DESCRIPTION:
Although use of marijuana is widespread, little research has focused on the treatment of marijuana use disorders or on predictors of relapse. Although several factors contributing to relapse have been explored in other dependencies (i.e., alcohol, cocaine), little research has focused on drug cue-related or stress-induced relapse in marijuana-dependent individuals. Cue reactivity is a construct measured in a laboratory procedure where an individual's subjective, behavioral, and physiological responses are assessed following exposure to drug-related environmental cues or stressors. Investigating the effects of drug-related environmental cues and stress in marijuana-dependent individuals will be useful in guiding treatment development.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Methods (DSM)-IV Criteria for Marijuana Dependence
* Between the ages of 18 and 65
* Must abstain from marijuana use the day of testing and other drug use three days prior to testing

Exclusion Criteria:

* Must not be taking any psychoactive medication, or medication that alters the hypothalamic pituitary adrenal (HPA) Axis functioning
* Must not be taking any medications that alter heart rate or skin conductance monitoring
* Cannot meet criteria for current major Axis I disorder (may alter response to stress)
* Cannot be morbidly obese (Body Mass Index >39)
* Cannot meet current abuse or dependence criteria of other substances in past 90 days
* Must not have a medical condition that impacts HPA functioning (Hypertension, chronic pain, Addison's disease)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee L McRae, PharmD, BCPP, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited primarily through community advertisements between January 2008 and June 2009.
Groups:
- Stress: Participants assigned to this group are required to complete the Trier Social Stress Task, which involves delivering a 5-minute speech and performing a 5-minute math problem in front of an audience. They then complete a cue exposure session involving both neutral and marijuana-related cues.
- No Stress: Participants assigned to this group are required to read magazines for ten minutes. They then complete a cue exposure session involving both neutral and marijuana-related cues.
Period: Overall Study
Arm/Group | Stress | No Stress
Started | 45 | 42
Completed | 45 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stress | No Stress | Total
Number analyzed (Participants) | 45 | 42 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 42 | 87
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 29 | 29 | 58
Region of Enrollment [Number; unit: participants]
  United States | 45 | 42 | 87

OUTCOME MEASURES:

1. Primary Outcome: Subjective Craving of Marijuana
Description: Defined as the score on the Marijuana Craving Questionnaire (MCQ), range 7-84, higher scores indicate more craving
Time Frame: approx 2.5 hours (before, during and after exposure to stressor condition as well as exposure to neutral and marijuana-associated cues).
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Stress | No Stress
Number analyzed (Participants) | 45 | 42
Scores on a Scale | 50.5 (1.6) | 52.3 (1.6)

2. Secondary Outcome: Physiological Assessments: Serum Cortisol, ACTH, BP, HR, and GSR
Time Frame: ~ 2.5 hours (before, during and after exposure to stressor condition as well as exposure to neutral and marijuana-associated cues).
Reporting Status: Not Posted

3. Secondary Outcome: Feelings of Stress/Anxiety as Measured by the State-Trait Inventory (STAI)
Time Frame: ~2 hours
Reporting Status: Not Posted

4. Secondary Outcome: Current Mood as Assessed by the Mood Form
Time Frame: ~2 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Stress | No Stress
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/42
Other Adverse Events (participants affected / at risk) | 0/45 | 0/42

LIMITATIONS AND CAVEATS:
A control group of non-marijuana dependent individuals was not included, which may have provided further insight into the interactions of stress and cues both in the presence and absence of addiction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No